CLINICAL TRIAL: NCT06671054
Title: A Randomized, Double Blind, Placebo-controlled, Dose Response, Phase II, Multicentre Trial to Evaluate the Efficacy and Safety of Oral AP1189 Administered at the Doses of 40, 70, or 100 mg for 12 Weeks in Combination With Methotrexate, in DMARD-naïve Participants With Early Rheumatoid Arthritis and Active Inflammation.
Brief Title: A Dose Response Study to Evaluate the Efficacy and Safety of Oral AP1189 Administered in Disease-Modifying Anti-Rheumatic Drug (DMARD) naïve Participants Participants With Early Rheumatoid Arthritis
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SynAct Pharma Aps (Industry)
Collaborators: NBCD A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SynAct-CS008
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-10

CONDITIONS: Rheumatoid Arthritis (RA)
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — N-(3-(1-(2-nitrophenyl)-1H-pyrrol-2-yl)allylidenamino)guanidine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- AP1189 40 mg (Experimental): 12 weeks daily treatment of oral AP1189 40 mg as add-on to Methotrexate (MTX)
  Interventions: Drug: AP1189, 40 mg
- AP1189 70 mg (Experimental): 12 weeks daily treatment of oral AP1189 70 mg as add-on to Methotrexate (MTX)
  Interventions: Drug: AP1189, 70 mg
- AP1189 100 mg (Experimental): 12 weeks daily treatment of oral AP1189 100 mg as add-on to Methotrexate (MTX)
  Interventions: Drug: AP1189, 100 mg
- Placebo (Experimental): 12 weeks daily treatment of oral AP1189 matching placebo as add-on to Methotrexate (MTX)
  Interventions: Drug: AP1189 matching placebo

INTERVENTIONS:
Drug: AP1189, 40 mg — AP1189 tablets for oral use
  Arms: AP1189 40 mg
Drug: AP1189, 70 mg — AP1189 tablets for oral use
  Arms: AP1189 70 mg
Drug: AP1189, 100 mg — AP1189 tablets for oral use
  Arms: AP1189 100 mg
Drug: AP1189 matching placebo — AP1189 tablets for oral use
  Arms: Placebo

SUMMARY:
The study is a randomized, double blind, placebo-controlled, dose response, phase II, multicentre trial to evaluate the efficacy and safety of oral AP1189 administered at the doses of 40, 70, or 100 mg for 12 weeks in combination with methotrexate, in DMARD-naïve participants with early rheumatoid arthritis and active inflammation.

DETAILED DESCRIPTION:
The purpose of the trial is to evaluate the efficacy, safety and tolerability of 12 weeks daily treatment of oral AP1189 at the doses of 40, 70, or 100 mg in combination with oral MTX compared to oral MTX alone.

The aim is to have 240 participants randomized to one of the 4 treatment groups, in a 1:1:1:1 ratio and treated with both AP1189/Placebo and MTX.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent obtained before undergoing any trial-specific procedure.
* Participants with definite RA diagnosis according to the 2010 American College of Rheumatology (ACR)/European League Against Rheumatism (EULAR) classification criteria.
* Disease duration no longer than 6 months from diagnosis at the time of Baseline Visit and with a history of RA symptoms which does not exceed 18 months.
* Participants must be naïve to any Disease-modifying anti-rheumatic drugs (DMARDs)
* Participants with at least 6/68 tender and 6/66 swollen joints at Screening Visit and Baseline.
* Participants with "high" disease activity as documented by a Disease Activity Score 28 (DAS28) (C-Reactive Protein - CRP) index score > 5.1 at screening, and Clinical disease activity index (CDAI) >22 at Screening Visit and Baseline.
* Participants with serum high sensitive C-Reactive Protein (hsCRP) ≥3 mg/L at the time of screening.
* Participants positive for serum rheumatoid factor (RF), AND/OR anti-cyclic citrullinated peptide antibodies (anti-CCP). If seronegative RA, hsCRP ≥6 mg/L at the time of screening.
* Willing and able to comply with the scheduled study visits, the treatment plan, and all study procedures.
* Females of childbearing potential must have a negative pregnancy test at screening and again at baseline.
* Sexually active female participants of childbearing potential and male participants are excluded if not practicing two different methods of birth control with their partner during the study and for 90 days after the last dose of study drug or who will not remain abstinent during the study and for 90 days after the last dose.

Exclusion Criteria:

* Functional class IV of Global Functional Status in RA, as defined by the ACR Classification.
* Rheumatic autoimmune disease other than RA, i.e. systemic lupus erythematosus, mixed connective tissue disease, scleroderma, polymyositis, or significant systemic involvement secondary to RA.
* Current inflammatory joint disease other than RA.
* Non-inflammatory type of musculoskeletal condition that in the Investigator's opinion is symptomatic and/or severe enough to interfere with the subject's primary diagnosis of RA or the evaluation of the effect of the study drug.
* Gastrointestinal diseases known to interfere with the absorption or excretion of medications.
* Severe, progressive, or uncontrolled renal, hepatic, hematologic, gastrointestinal, metabolic, endocrine, pulmonary, cardiac or neurologic disease.
* Malignancy active during the 12 months preceding the Screening Visit.
* Acute hepatitis, chronic hepatitis, or detection of any unexplained elevation of serum ALT or AST greater than 1.5-fold ULN, at least twice in the 6 months before the Screening Visit) or HIV infection.
* History of alcohol or drug abuse during the 12 months preceding the Screening Visit.
* Vaccination with live vaccines during the 6 weeks preceding the Screening Visit.
* Haemoglobin <9 g/dL or Haematocrit <30% at the Screening Visit
* White blood cell (WBC) count <3.0 x 109/L at the Screening Visit.
* Absolute neutrophil count <1.2 x 109/L at the Screening Visit.
* Platelet count <100 x 109/L at the Screening Visit.
* Serum alkaline-phosphatase, or gamma-glutamyl-transferase greater than 3-fold ULN; alanine aminotransferase, or aspartate aminotransferase, or total bilirubin greater than 2-fold ULN At the Screening Visit.
* Estimated creatinine clearance less than 45 mL/min/1.73 m2 (MDRD) at the Screening Visit.
* 12-lead electrocardiogram (ECG) with abnormal clinically significant findings, as judged by the Investigator, at the Screening Visit.
* Positive QuantiFERON-in-Tube test (QFG-IT).
* Use of hydroxychloroquine during the 30 weeks preceding the Screening Visit.
* Treatment with any systemic or intraarticular corticosteroid within 6 weeks before the Screening Visit.
* Intermittent use of nonsteroidal anti-inflammatory drugs (NSAIDs). Use of NSAIDs is allowed if used in a stable dose regimen for at least 4 weeks prior to the Screening Visit.
* Use of other investigational drugs/treatments, or enrolment in a clinical trial during the 6 months preceding the Screening Visit.
* Any other clinically relevant disease and condition that, in the opinion of the Investigator, may jeopardize efficacy or safety assessments or may compromise the subject's safety during trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Disease Activity Score 28 (DAS28)-C-Reactive Protein (CRP) | Week 12
  Absolute change from baseline in DAS28-CRP at Week 12

CONTACTS AND LOCATIONS:
Locations (11):
- United States (3):
  - Nouvelle Clinical Research LLC, Cutler Bay, Florida
  - Millennium Medical Research LLC, Miami, Florida
  - Altoona Center for Clinical Research, Duncansville, Pennsylvania
- Bulgaria (2):
  - Diagnostic Consultative Center Aleksandrovska, Sofia
  - Medical Center Tera Medico, Vratsa
- Sanos Clinic Herlev, Herlev, Denmark
- IMSP Spitalul Clinic Municipal "Sfanta Treime", Chisinau, Moldova
- Poland (4):
  - M2Mmed, Chorzów
  - Vita Longa Sp. z o. o., Katowice
  - Medyczne Centrum Hetmańska, Poznan
  - DC-MED Michal Kowalski S.K., Swidnica

IPD SHARING:
Plan to Share IPD: No